CLINICAL TRIAL: NCT06626555
Title: Pilot, Randomized, Open-Label, Non-Active Comparator Controlled Clinical Trial to Evaluate the Effects of Letermovir Prophylaxis on T-cell Immune Activation in Participants With Treated HIV-1 Infection
Brief Title: Clinical Trial to Evaluate the Effects of Letermovir Prophylaxis on T-cell Immune Activation in Participants With Treated HIV-1 Infection
Acronym: PROACTIV
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 125096; 2020-000288-22 (EudraCT Number)
Record Dates: First submitted 2024-08-14; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: HIV
MeSH Terms: interventions — letermovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Letermovir (Experimental): Letermovir 480mg PO once daily
  Interventions: Drug: Letermovir
- Standard of Care (No Intervention): Standard of care - No intervention

INTERVENTIONS:
Drug: Letermovir — Letermovir 480mg PO once daily
  Arms: Letermovir

SUMMARY:
People living with HIV (PLWH), even with an undetectable viral load (VL) on antiretroviral treatment (ART), develop health conditions, such as heart disease, diabetes, various cancers, and conditions that can affect the brain, more commonly than the general population.

These conditions occur earlier in PLWH compared to HIV negative individuals with similar lifestyles. Ongoing inflammation in the body despite antiretroviral therapy is thought to be contributing to the development of these conditions that can affect healthy ageing in PLWH.

Cytomegalovirus (CMV) is a very common infection in PLWH and is an important driver of inflammation in the body that can affect the function of the immune immune cells in the body (defense system) causing unwanted activation and damage of the gut making it more leaky. A drug with potent activity against CMV called valganciclovir has previously shown to reduce this potentially damaging inflammation in the body.

In this study, the investigators want to investigate if a new drug called Letermovir, in combination with HIV treatment, will prevent CMV from replicating (multiplying), and thereby reduce inflammation in the body. Letermovir has received approval to prevent CMV from multiplying in patients receiving bone marrow transplants. It has been shown to have a more favourable side-effect profile compared to other available drugs and is predicted to interact little with anti-HIV drugs.

The aim of this study is to find out if the letermovir is safe and effective in reducing CMV related immune activation and inflammation PLWH. These findings will be used to help us design larger studies to identify individuals who would benefit most from this treatment to prevent the development of health conditions that can affect their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Is HIV-1 antibody positive with a plasma HIV-1 RNA ≤50 copies/mL for greater than 12 months
* ≥50 years of age of any gender
* Females of childbearing potential who agree to avoid pregnancy for the duration of the trial and follow methods of contraception as detailed in section 7.1
* Has a nadir CD4 of ≤200 cells/mm3 prior to screening
* Has been on antiretroviral therapy for ≥ 6 months
* Has documented CMV IgG seropositivity within one year of trial screening
* Has an undetectable (≤168 international units/mL) CMV Deoxyribonucleic acid (DNA) within 14 days prior to randomisation
* Laboratory parameters are not clinically significant as determined by the investigator
* The participant (or legally acceptable representative, if applicable) has provided written informed consent for the trial and Future Biomedical Research

Exclusion Criteria:

* Is HIV-1 antibody positive with a plasma HIV-1 RNA ≤50 copies/mL for greater than 12 months
* ≥50 years of age of any gender
* Females of childbearing potential who agree to avoid pregnancy for the duration of the trial and follow methods of contraception as detailed in section 7.1
* Has a nadir CD4 of ≤200 cells/mm3 prior to screening
* Has been on antiretroviral therapy for ≥ 6 months
* Has documented CMV IgG seropositivity within one year of trial screening
* Has an undetectable (≤168 international units/mL) CMV Deoxyribonucleic acid (DNA) within 14 days prior to randomisation
* Laboratory parameters are not clinically significant as determined by the investigator
* The participant (or legally acceptable representative, if applicable) has provided written informed consent for the trial and Future Biomedical Research

Main Exclusion criteria:

* Has a history of ulcerative colitis or Crohn's disease or active colitis within 6 months prior to randomisation
* Has a history of CMV end-organ disease within 6 months prior to randomisation
* Has significant hypersensitivity or other contraindication to any of the components of the trial drug as described in the SmPC
* Has a detectable HCV RNA or hepatitis B surface antigen (HBsAg) within 90 days prior to randomisation
* Has a history of malignancy ≤5 years prior to signing informed consent
* Is pregnant or expecting to conceive, is breastfeeding, or plans to breastfeed from the time of consent through 90 days after the last dose of trial therapy
* Has received within 7 days prior to screening any of the following: ganciclovir; valganciclovir; foscarnet; acyclovir (≥ 3200 mg PO per day or ≥25 mg/kg IV per day); valaciclovir (≥3000 mg PO per day) or famciclovir (≥1500 mg PO per day).
* Has used systemic immunosuppressive therapy or immune modulators within 30 days prior to treatment in this trial or is anticipated to need them during the trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in activation in global CD8 T cells in response to letermovir. | Baseline, weeks 4, 8, 12, 16 and 24
  To assess the effect of CMV replication inhibition with letermovir on activated (HLADR+CD38+) CD8 T cell percentage using flow cytometry analysis at specified time frames.
  Measurement: Measured by flow cytometric analysis.

SECONDARY OUTCOMES:
Quantitative analysis of T cell subsets/detailed phenotypic profile will be performed as part of the exploratory analysis | Baseline, weeks 12 and 24
  Quantitative analysis of T cell subsets/detailed phenotypic profile will be performed as part of the exploratory analysis
Characterization of NK profile and function in response to Letermovir | Baseline, weeks 4, 8, 12, 16 and 24
  To assess the effect of CMV replication inhibition with letermovir on NK cell phenotype and cytokine production (IFN-g/TNF) via flow cytometry.
  Measurement: Measured by flow cytometric analysis.
High resolution characterization of cells that fall between the innate and adaptive responses | Baseline, weeks 12 and 24
  To assess the effect of CMV replication inhibition with letermovir on NK-like cells (CD56+CD3+) at specified time points.
  Measurement: Measured by flow cytometric analysis.
Determine the extent of CMV and HIV replication in the gut of HIV-positive individuals and how impacted by intervention | Baseline, weeks 12 and 24
  To assess CMV DNA and HIV RNA in gut biopsies and the effect of intervention. Measurement: Measured by quantitative PCR analysis and in situ hybridisation.
Assessment of integrity of the intestinal barrier and how impacted by intervention | Baseline, weeks 12 and 24
  To assess the influence of CMV replication inhibition with letermovir on intestinal barrier integrity in gut biopsies.
  Measurement: Measured by immunohistochemistry of biopsy samples for zonula occludens-1 (ZO-1).
Assessment of markers of systemic inflammation and how impacted by intervention | Baseline, weeks 4, 8, 12, 16 and 24
  To assess the influence of CMV replication inhibition with letermovir on inflammatory cytokines/chemokines (IL-1, IL-6, IP10, TNF-a), sTNFRII, microbial products/activation (LPS, sCD14, CRP), intestinal damage marker (iFABP), vascular dysfunction markers (sICAM-1, sVCAM-1) in the blood of people with HIV.
  Measurement: Measured by ELISA.

OTHER OUTCOMES:
Higher resolution analysis of specific responses to peptide level and how impacted by intervention | Baseline, weeks 4, 8, 12, 16 and 24
  To assess the influence of letermovir on CMV and HIV-specific T cell responses to peptide stimulation via multiparameter intracellular cytokine staining. Expression of cytokines, such as IFN-γ, TNF and IL-2, and activation markers will be measured via flow cytometry in conjunction with established phenotypic and memory markers.
  Measurement: Measured by flow cytometric analysis
Standard molecular analyses of proviral and HIV transcript quantitation, both surrogate markers of persistent infection | Baseline, weeks 4, 8, 12, 16 and 24
  To assess the influence of CMV replication inhibition with letermovir on HIV DNA and Cell-associated RNA Measure: Measured by quantitative real-time PCR and droplet digital PCR (ddPCR).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hunt PW, Martin JN, Sinclair E, Epling L, Teague J, Jacobson MA, Tracy RP, Corey L, Deeks SG. Valganciclovir reduces T cell activation in HIV-infected individuals with incomplete CD4+ T cell recovery on antiretroviral therapy. J Infect Dis. 2011 May 15;203(10):1474-83. doi: 10.1093/infdis/jir060. PMID 21502083
- [Background] Bradley T, Peppa D, Pedroza-Pacheco I, Li D, Cain DW, Henao R, Venkat V, Hora B, Chen Y, Vandergrift NA, Overman RG, Edwards RW, Woods CW, Tomaras GD, Ferrari G, Ginsburg GS, Connors M, Cohen MS, Moody MA, Borrow P, Haynes BF. RAB11FIP5 Expression and Altered Natural Killer Cell Function Are Associated with Induction of HIV Broadly Neutralizing Antibody Responses. Cell. 2018 Oct 4;175(2):387-399.e17. doi: 10.1016/j.cell.2018.08.064. Epub 2018 Sep 27. PMID 30270043
- [Background] Thornhill JP, Pace M, Martin GE, Hoare J, Peake S, Herrera C, Phetsouphanh C, Meyerowitz J, Hopkins E, Brown H, Dunn P, Olejniczak N, Willberg C, Klenerman P, Goldin R, Fox J, Fidler S, Frater J; CHERUB investigators. CD32 expressing doublets in HIV-infected gut-associated lymphoid tissue are associated with a T follicular helper cell phenotype. Mucosal Immunol. 2019 Sep;12(5):1212-1219. doi: 10.1038/s41385-019-0180-2. Epub 2019 Jun 25. PMID 31239514
- [Background] Amir el-AD, Davis KL, Tadmor MD, Simonds EF, Levine JH, Bendall SC, Shenfeld DK, Krishnaswamy S, Nolan GP, Pe'er D. viSNE enables visualization of high dimensional single-cell data and reveals phenotypic heterogeneity of leukemia. Nat Biotechnol. 2013 Jun;31(6):545-52. doi: 10.1038/nbt.2594. Epub 2013 May 19. PMID 23685480
- [Background] Levine JH, Simonds EF, Bendall SC, Davis KL, Amir el-AD, Tadmor MD, Litvin O, Fienberg HG, Jager A, Zunder ER, Finck R, Gedman AL, Radtke I, Downing JR, Pe'er D, Nolan GP. Data-Driven Phenotypic Dissection of AML Reveals Progenitor-like Cells that Correlate with Prognosis. Cell. 2015 Jul 2;162(1):184-97. doi: 10.1016/j.cell.2015.05.047. Epub 2015 Jun 18. PMID 26095251
- [Background] Peppa D, Pedroza-Pacheco I, Pellegrino P, Williams I, Maini MK, Borrow P. Adaptive Reconfiguration of Natural Killer Cells in HIV-1 Infection. Front Immunol. 2018 Mar 16;9:474. doi: 10.3389/fimmu.2018.00474. eCollection 2018. PMID 29616021
- [Background] Gupta RK, Abdul-Jawad S, McCoy LE, Mok HP, Peppa D, Salgado M, Martinez-Picado J, Nijhuis M, Wensing AMJ, Lee H, Grant P, Nastouli E, Lambert J, Pace M, Salasc F, Monit C, Innes AJ, Muir L, Waters L, Frater J, Lever AML, Edwards SG, Gabriel IH, Olavarria E. HIV-1 remission following CCR5Delta32/Delta32 haematopoietic stem-cell transplantation. Nature. 2019 Apr;568(7751):244-248. doi: 10.1038/s41586-019-1027-4. Epub 2019 Mar 5. PMID 30836379
- [Background] Gupta RK, Peppa D, Hill AL, Galvez C, Salgado M, Pace M, McCoy LE, Griffith SA, Thornhill J, Alrubayyi A, Huyveneers LEP, Nastouli E, Grant P, Edwards SG, Innes AJ, Frater J, Nijhuis M, Wensing AMJ, Martinez-Picado J, Olavarria E. Evidence for HIV-1 cure after CCR5Delta32/Delta32 allogeneic haemopoietic stem-cell transplantation 30 months post analytical treatment interruption: a case report. Lancet HIV. 2020 May;7(5):e340-e347. doi: 10.1016/S2352-3018(20)30069-2. Epub 2020 Mar 10. PMID 32169158
- [Background] Alrubayyi A, Gea-Mallorqui E, Touizer E, Hameiri-Bowen D, Kopycinski J, Charlton B, Fisher-Pearson N, Muir L, Rosa A, Roustan C, Earl C, Cherepanov P, Pellegrino P, Waters L, Burns F, Kinloch S, Dong T, Dorrell L, Rowland-Jones S, McCoy LE, Peppa D. Characterization of humoral and SARS-CoV-2 specific T cell responses in people living with HIV. Nat Commun. 2021 Oct 5;12(1):5839. doi: 10.1038/s41467-021-26137-7. PMID 34611163